CLINICAL TRIAL: NCT01251276
Title: A Study to Estimate the Immune Response Following a Challenge Dose in Adults (≥50 Years Old) Vaccinated With a Primary Series of an Hepatitis B Vaccine
Brief Title: Hepatitis B Challenge Dose in Adults (V232-059-10)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V232-059-10; rHB01C (Other: MCMVaccBV (SPMSD) Protocol Number); 2006-003649-18 (EudraCT Number)
Record Dates: First submitted 2010-11-23; First posted 2010-12-01 (Estimated); Results first posted 2017-08-28 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-08

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — Hepatitis B Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Modified Process Hepatitis B Vaccine in Base Study (Experimental): Participants who received 3 doses of Modified Process Hepatitis B Vaccine in the Base Study were eligible to receive a single challenge dose of Modified Process Hepatitis B Vaccine on Day 1 of the Challenge Dose Study
  Interventions: Biological: Modified Process Hepatitis B Vaccine
- ENGERIX-B™ Vaccine in Base Study (Experimental): Participants who received 3 doses of ENGERIX-B™ vaccine in the Base Study were eligible to receive a single challenge dose of Modified Process Hepatitis B Vaccine on Day 1 of the Challenge Dose Study
  Interventions: Biological: Modified Process Hepatitis B Vaccine

INTERVENTIONS:
Biological: Modified Process Hepatitis B Vaccine — Modified Process Hepatitis B Vaccine given IM (intramuscular) as a single 1.0 mL (10 mcg) challenge dose on Day 1 of the Challenge Dose Study
  Other Names: HBVaxPro

SUMMARY:
The purpose of this trial is to describe the Seroprotection Rate (SPR) at least 2 years following completion of a primary series with a hepatitis B vaccine (Base Study V232-059, NCT00440531) and 1 month following a challenge dose with a Modified Process Hepatitis B vaccine.

ELIGIBILITY:
Inclusion Criteria:

* In general good health based on a medical history.
* Received 3 doses of an Hepatitis B vaccine in Base Study V232-059, NCT00440531 at least 2 years prior to enrollment in this study.

Exclusion Criteria:

* Known history of previous Hepatitis B infection.
* History of vaccination with any Hepatitis B vaccine within the last 2 years.
* History of febrile illness.
* Known or suspected hypersensitivity to any component of HBVaxPro.
* Receipt of medication / vaccine that may interfere with study assessments.
* Known or suspected immune impairment.
* Pregnant women and nursing mothers.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2010-11-30 (Actual); Primary Completion 2011-04-12 (Actual); Study Completion 2011-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Sharma R, Ahlm C, Ostergaard L, Dowell A, Tran C, Thomas S, Eymin C. Persistence of immunity in healthy adults aged >/= 50 years primed with a hepatitis B vaccine 3 years previously. Hum Vaccin Immunother. 2015;11(7):1709-16. doi: 10.1080/21645515.2015.1019187. PMID 25996838

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 296 participants were eligible for the challenge-dose study and 204 were enrolled
Pre-assignment Details: Study participants received 3 doses of Modified Process Hepatitis B Vaccine or ENGERIX-B™ vaccine in the Base Study (V232-059, NCT00440531). Two years after completion of the Base Study vaccinations, participants were eligible to receive one challenge dose of Modified Process Hepatitis B Vaccine on Day 1 of the Challenge Dose Study.
Groups:
- Modified Process Hepatitis B Vaccine in Base Study: Participants who received 3 doses of Modified Process Hepatitis B Vaccine in the Base Study received a single challenge dose of Modified Process Hepatitis B Vaccine on Day 1 of the Challenge Dose Study
- ENGERIX-B™ Vaccine in Base Study: Participants who received 3 doses of ENGERIX-B™ vaccine in the Base Study received a single challenge dose of Modified Process Hepatitis B Vaccine on Day 1 of the Challenge Dose Study
Period: Overall Study
Arm/Group | Modified Process Hepatitis B Vaccine in Base Study | ENGERIX-B™ Vaccine in Base Study
Started | 96 (Not all Base Study completers enrolled in the Challenge Dose Study) | 108 (Not all Base Study completers enrolled in the Challenge Dose Study)
Vaccinated | 96 | 108
Completed | 95 | 107
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled and vaccinated participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Modified Process Hepatitis B Vaccine in Base Study | ENGERIX-B™ Vaccine in Base Study | Total
Number analyzed (Participants) | 96 | 108 | 204
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at the time of challenge dose
  Years | 63.8 (7.3) | 63.6 (6.7) | 63.7 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 63 | 111
  Male | 48 | 45 | 93

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Seroresponders Before and After the Challenge Vaccination
Description: A seroresponder was a participant with an anti-hepatitis B surface antibody titer >=10 milli Merck U/mL. The percentage of seroresponders was assessed before and after the challenge dose.
Time Frame: Predose (Day 1) and 1 month after challenge dose (Month 1)
Population: Vaccinated participants with immunogenicity results, excluding those with protocol violations that might interfere with the immunogenicity evaluation
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Modified Process Hepatitis B Vaccine in Base Study | ENGERIX-B™ Vaccine in Base Study
Number analyzed (Participants) | 88 | 103
Percentage of participants
  Predose (Day 1); n=88, 102 | 45.5 [34.8 to 56.4] | 58.8 [48.6 to 68.5]
  Postdose (Month 1); n=88, 103 | 85.2 [76.1 to 91.9] | 88.3 [80.5 to 93.8]

2. Secondary Outcome: Percentage of Participants With One or More Adverse Experiences
Description: An adverse experience is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the sponsor's product, whether or not considered related to the use of the product. Any worsening of a preexisting condition which is temporally associated with the use of the sponsor's product, is also an adverse experience. The percentage of participants with one or more adverse experiences was assessed.
Time Frame: Up to Day 15 after challenge dose
Population: Participants who received a challenge dose and had safety follow-up
Measure: Number; unit: Percentage of participants
Arm/Group | Modified Process Hepatitis B Vaccine in Base Study | ENGERIX-B™ Vaccine in Base Study
Number analyzed (Participants) | 96 | 107
Percentage of participants | 39.6 | 45.8

3. Secondary Outcome: Percentage of Participants Who Discontinued the Study Due to an Adverse Experience
Description: The percentage of participants who discontinued the study due to an adverse experience was assessed.
Time Frame: Up to Month 7
Population: Participants who received a challenge dose and had safety follow-up
Measure: Number; unit: Percentage of participants
Arm/Group | Modified Process Hepatitis B Vaccine in Base Study | ENGERIX-B™ Vaccine in Base Study
Number analyzed (Participants) | 96 | 107
Percentage of participants | 0 | 0

4. Secondary Outcome: Percentage of Participants With One or More Injection-site Adverse Experiences
Description: The percentage of participants with one or more injection-site adverse experiences was assessed.
Time Frame: Up to Day 15 after challenge dose
Population: Participants who received a challenge dose and had safety follow-up
Measure: Number; unit: Percentage of participants
Arm/Group | Modified Process Hepatitis B Vaccine in Base Study | ENGERIX-B™ Vaccine in Base Study
Number analyzed (Participants) | 96 | 107
Percentage of participants | 35.4 | 29.9

5. Secondary Outcome: Percentage of Participants With One or More Systemic Adverse Experiences
Description: The percentage of participants with one or more systemic adverse experiences was assessed.
Time Frame: Up to Day 15 after challenge dose
Population: Participants who received a challenge dose and had safety follow-up
Measure: Number; unit: Percentage of participants
Arm/Group | Modified Process Hepatitis B Vaccine in Base Study | ENGERIX-B™ Vaccine in Base Study
Number analyzed (Participants) | 96 | 107
Percentage of participants | 16.7 | 28.0

6. Secondary Outcome: Percentage of Participants With One or More Serious Adverse Experiences
Description: A serious adverse experience is an adverse experience that results in death, is life threatening, results in persistent or significant disability or incapacity, results in or prolongs a hospitalization, is a congenital anomaly or birth defect, is a cancer, or may jeopardize the participant and may require medical or surgical intervention. The percentage of participants with one or more serious adverse experiences was assessed.
Time Frame: Up to Month 1 after challenge dose
Population: Participants who received a challenge dose and had safety follow-up
Measure: Number; unit: Percentage of participants
Arm/Group | Modified Process Hepatitis B Vaccine in Base Study | ENGERIX-B™ Vaccine in Base Study
Number analyzed (Participants) | 96 | 107
Percentage of participants | 0 | 0.9

ADVERSE EVENTS:
Time Frame: All adverse events: up to Day 15 after the challenge dose; serious adverse events: up to 1 month after the challenge dose
Description: The Safety Analysis Set included participants who received the challenge dose vaccination and had safety follow-up
Arm/Group | Modified Process Hepatitis B Vaccine in Base Study | ENGERIX-B™ Vaccine in Base Study
Serious Adverse Events (participants affected / at risk) | 0/96 | 1/107
Other Adverse Events (participants affected / at risk) | 34/96 | 30/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Modified Process Hepatitis B Vaccine in Base Study (N=96) | ENGERIX-B™ Vaccine in Base Study (N=107)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Modified Process Hepatitis B Vaccine in Base Study (N=96) | ENGERIX-B™ Vaccine in Base Study (N=107)
Injection-site erythema (General disorders) | 7 (7) | 5 (5)
Injection-site pain (General disorders) | 31 (31) | 27 (27)
Injection-site swelling (General disorders) | 7 (7) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study sixty (60) days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.